CLINICAL TRIAL: NCT02192918
Title: Pilot Investigation of Behavioral Alternatives to Indoor Tanning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Sherry Pagoto, Associate Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R21CA161576-01A1 (NIH)
Record Dates: First submitted 2014-06-09; First posted 2014-07-17 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Airbrush (Experimental): Participants will receive the American Academy of Dermatology Sun Smart pamphlet at the baseline session. It has brief tips for reducing skin cancer risk, but does not mention sunless tanning or relaxation activities. Participants will also complete 4 airbrush tan sessions, once every two weeks, over the course of 2 months. Participants will receive access to one of each of the following after the 6-month assessment at no cost: massage, pedicure, yoga class, and dance class. Participants will schedule these activities on their own and the study staff will arrange for payment for the appointment.
  Interventions: Behavioral: Airbrush
- Airbrush Plus (Experimental): Participants will receive the American Academy of Dermatology Sun Smart pamphlet at the baseline session. It has brief tips for reducing skin cancer risk, but does not mention sunless tanning or relaxation activities. Participants will also complete 4 airbrush tan sessions, once every two weeks, over the course of 2 months. Additionally, they may choose 8 sessions, 1 per week, of the following activities at no cost: massage, pedicure, yoga class, or dance class. These activities are being given as healthy alternatives to the relaxation sensation of indoor tanning.
  Interventions: Behavioral: Airbrush Plus
- Delayed Airbrush Plus (Active Comparator): Participants will receive the American Academy of Dermatology Sun Smart pamphlet at the baseline session. It has brief tips for reducing skin cancer risk, but does not mention sunless tanning or relaxation activities. Participants will also receive access to one of each of the following after the 6-month assessment at no cost: airbrush tan, massage, pedicure, yoga class, and dance class.
  Interventions: Behavioral: Delayed Airbrush

INTERVENTIONS:
Behavioral: Airbrush — The American Academy of Dermatology Sun Smart pamphlet will be given at the baseline session. It has brief tips for reducing skin cancer risk, but does not mention sunless tanning or relaxation activities. Participants in the airbrush condition will receive 4 airbrush tan sessions, once every two weeks, over the course of 2 months.
  Arms: Airbrush
Behavioral: Airbrush Plus — The American Academy of Dermatology Sun Smart pamphlet will be given at the baseline session. It has brief tips for reducing skin cancer risk, but does not mention sunless tanning or relaxation activities. Participants will complete 4 airbrush tan sessions, once every two weeks, over the course of 2 months. Additionally, they may choose 8 sessions, 1 per week, of the following activities at no cost: massage, pedicure, yoga class, or dance class.
  Arms: Airbrush Plus
Behavioral: Delayed Airbrush — The American Academy of Dermatology Sun Smart pamphlet will be given at the baseline session. It has brief tips for reducing skin cancer risk, but does not mention sunless tanning or relaxation activities. Participants will receive access to one of each of the following after the 6-month assessment at no cost: airbrush tan, massage, pedicure, yoga class, and dance class
  Arms: Delayed Airbrush Plus

SUMMARY:
The goal of this research is to develop and test the feasibility of an intervention that stimulates uptake of healthy alternatives to tanning by providing free access to them for a limited time. Free access gives participants a low-risk opportunity to try something new that is consistent with their motivations. Free access also allows them to experience the reinforcing properties of the alternatives which could prime continued use after the free trial period. The objective of the present study is to determine the feasibility and short-term efficacy of providing free alternatives to indoor tanners in an effort to "nudge" them to switch from indoor tanning to healthy alternatives.

DETAILED DESCRIPTION:
Melanoma is the second most common cancer diagnosed in young women and is responsible for nearly 8,000 US deaths per year. Exposure to ultraviolet radiation (UVR) increases risk for melanoma. The International Agency for Research on Cancer assigned indoor tanning (IT; use of tanning beds or booths), as a class 1 carcinogen joining arsenic, asbestos, and mustard gas. Unfortunately, interventions educating tanners about the risks have not been very effective. Many tanners are more motivated by the immediate consequences of tanning than the delayed consequence of possibly getting cancer. Research shows the primary motivation for indoor tanning is to improve physical appearance, but a secondary motivation is stress reduction. Behavioral economics theory suggests that the rate of a behavior depends on 1) the reinforcing value of that behavior relative to alternatives, 2) the cost of engaging in the behavior relative to alternatives, and 3) the availability of the behavior relative to alternatives. The purpose of the present study is to determine whether exposure to healthy alternatives changes the behavior of indoor tanners. The investigators will randomize tanners to conditions differing in physical appearance and stress reduction alternatives to determine whether they can get their motivational needs met in healthier ways.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 16-65
* Report minimum of 10 indoor tanning visits in the last year with intentions to continue

Exclusion Criteria:

* Ages <16 or >65
* Pregnant, breastfeeding, or planning to become pregnant during the study period
* Reporting less than 10 indoor tanning visits per year
* No intention to continue indoor tanning
* Using sunless tanning more than once in the last year and ever in the last 3 months
* Physically limited to do yoga or dance classes
* DHA allergy
* Inability to consent
* Prisoners

Ages: 16 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Satisfaction | up to 12 months
  A measure of satisfaction will be assessed for each alternative visit on a scale of 1-10 immediately after each activity is completed. Visits occur between baseline and 12 months of participation. Timing of visits depend on which condition is assigned.
Effort of alternatives | 6-month follow-up
  Perceived effort of alternatives will be discussed in a focus group setting.
Recruitment rate | baseline
  Total randomized and total screened out.
Retention | 12 month follow-up
  % sessions complete and total withdrawn from study

SECONDARY OUTCOMES:
abstinence | 2-month follow-up
  the percent of participants who abstained from indoor tanning.
abstinence | 3-month follow-up
  the percent of participants who abstained from indoor tanning.
abstinence | 6-month follow-up
  the percent of participants who abstained from indoor tanning.
abstinence | 12-month follow-up
  the percent of participants who abstained from indoor tanning.

OTHER OUTCOMES:
Cost of indoor tanning | 2-month follow-up
  Total amount spent on tanning since the previous assessment.
Cost of indoor tanning | 3-month follow-up
  Total amount spent on tanning since the previous assessment.
Cost of indoor tanning | 6-month follow-up
  Total amount spent on tanning since the previous assessment.
Cost of indoor tanning | 12-month follow-up
  Total amount spent on tanning since the previous assessment.
Stress Level | 2-month follow-up
  Perceived Stress Scale
Stress Level | 3-month follow-up
  Perceived Stress Scale
Stress Level | 6-month follow-up
  Perceived Stress Scale
Stress Level | 12-month follow-up
  Perceived Stress Scale
Attitudes | 3-month follow-up
  Indoor Tanning Attitude Scale and the same scale modified for each of the alternatives
Attitudes | 6-month follow-up
  Indoor Tanning Attitude Scale and the same scale modified for each of the alternatives
Attitudes | 12-month follow-up
  Indoor Tanning Attitude Scale and the same scale modified for each of the alternatives
Tanning Dependence | 2-month follow-up
  modified CAGE
Tanning Dependence | 3-month follow-up
  modified CAGE
Tanning Dependence | 6-month follow-up
  modified CAGE
Tanning Dependence | 12-month follow-up
  modified CAGE

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Pagoto, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States